CLINICAL TRIAL: NCT07043842
Title: Effects of Thoracic Mobility Exercises Combined With Scapular Stabilization Exercises on Pain, Range of Motion, Scapular Alignment, Postural Alignment and Quality of Life in Individuals With Subacromial Pain Syndrome
Brief Title: Effect of Thoracic Mobility Exercises Combined With Scapular Stabilization Exercises in Individuals With Subacromial Pain Syndrome
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Ankara Yildirim Beyazıt University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 16.01.2025-01/1119
Record Dates: First submitted 2025-06-21; First posted 2025-06-29 (Actual); Last update posted 2025-06-29 (Actual); Status verified 2025-06

CONDITIONS: Subacromial Pain Syndrome
Keywords: subacromial pain syndrome; scapular stabilization exercises; thoracic mobility exercises

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Treatment group (Experimental): This group consists of patients who will undergo shoulder circumference exercises and scapular stabilization exercises along with thoracic mobility exercises.
  Interventions: Other: Shoulder circumference exercises; Other: Scapular stabilization exercises; Other: Thoracic mobility exercises
- Control group (Active Comparator): This group consists of patients who will undergo shoulder circumference exercises and scapular stabilization exercises.
  Interventions: Other: Shoulder circumference exercises; Other: Scapular stabilization exercises

INTERVENTIONS:
Other: Shoulder circumference exercises — They are strengthening and stretching exercises that support the range of motion of the shoulder joint.
Other: Scapular stabilization exercises — Changes in the biomechanics of the scapula affect the function of the shoulder. Biomechanical correction will be attempted with these exercises aimed at correcting the posture of the scapula.
Other: Thoracic mobility exercises — Changes in the biomechanics of the thoracic spine affect the function of the shoulder. Biomechanical correction will be attempted with these exercises aimed at correcting the posture of the thoracic spine.
  Arms: Treatment group

SUMMARY:
The subject of this study is to examine the effects of thoracic mobility exercises combined with scapular stabilization exercises on pain, range of motion, scapular alignment, postural alignment and quality of life in individuals with subacromial pain syndrome.

The scapula assumes a role that is attached to the axial skeleton by atmospheric pressure and axioscapular muscles, and prepares the ground for the formation of wide range of motion in the shoulder complex. The scapulothoracic movement formed by the movement of the scapula on the thorax is provided not only by the function of the scapular muscles but also by the optimization of the thoracic muscles and posture.

Therefore, changes in the biomechanics of the thoracic spine and scapula affect the function of the shoulder. Therefore, we predict that the possible contributions of scapular stabilization and thoracic mobility exercises to scapular alignment and alignment in thoracic posture will further improve shoulder-related complaints.

DETAILED DESCRIPTION:
Subacromial pain syndrome is one of the most common causes of shoulder pain. Factors leading to rotator cuff pathology due to decreased subacromial space play a role in its development. Depending on the stage of Subacromial Pain Syndrome; edema and hemorrhage in subacromial tissues, pain and tenderness in the lateral shoulder, fibrosis in the glenohumeral capsule and subacromial bursa, tendonitis in the affected tendons, abrasion, ruptures or osteophytes may develop in tendons. Again depending on the stage; postural changes such as increased downward rotation and anterior tilt in the scapula, loss of active-passive range of motion, atrophy in the rotator cuff and deltoid muscles may be observed. These disorders cause imbalances that may prevent optimal scapulohumeral rhythm. Changes in the biomechanics of the thoracic spine and scapula affect the function of the shoulder. Extension of the thoracic spine is significantly limited in subacromial pain syndrome. The scapula can also assume a significantly increased anterior tilt, internal rotation, protraction and decreased upward rotation position. This situation indicates that interventions are needed to improve limited thoracic extension and altered scapular position that may affect shoulder joint motion and muscle strength in the rehabilitation of individuals with subacromial pain syndrome.

A study on young tennis players, including thoracic region mobility exercises, based on the idea that increased thoracic kyphosis reduces shoulder functional capacity, has yielded effective results in correcting sagittal thoracic curvature and increasing thoracic mobility. It also strongly increased glenohumeral internal and external rotation range of motion.

Throwing injuries to the shoulder joint often occur during shoulder external rotation. Therefore, an appropriate combination of thoracic, scapular and humeral motion during throwing is important to prevent such injuries. Thoracic extension increases scapular posterior tilt and external rotation during shoulder external rotation and decreases glenohumeral horizontal abduction, and also increases maximum shoulder external rotation. It has been shown that providing thoracic extension can contribute to reducing mechanical demands on the glenohumeral joint during activities such as throwing and can potentially reduce shoulder injuries. Restricting thoracic extension can reduce scapulothoracic movement and cause excessive glenohumeral joint movement, which can be a risk factor for shoulder injuries. The finding of a significant positive correlation between scapular posterior tilt and glenohumeral external rotation also provides an idea about the posture that should be adopted to reduce the risk of injury. Therefore, during shoulder movements, it is necessary to correct the posture of the thoracic spine in order to prevent the incompatibility of scapula and thorax movements due to posture. Based on this, it is expected that the study to be conducted will shed light on the rehabilitation of individuals with subacromial pain syndrome by demonstrating the effectiveness of thoracic mobility exercises.

ELIGIBILITY:
Inclusion Criteria:

* Volunteering to participate in the study
* Being between the ages of 18-60
* Being diagnosed with subacromial pain syndrome
* Having Stage I or Stage II subacromial pain syndrome according to Neer
* Having unilateral shoulder pain that limits activity for more than 6 weeks
* Having pain intensity over 3 according to VAS

Exclusion Criteria:

* Having cervical radiculopathy
* Having spinal deformities
* Having post-traumatic symptom onset
* Having a history of shoulder dislocation or fracture
* Having passive joint movement limitation (frozen shoulder)
* Having received steroid injections within the last 6 weeks
* Having degenerative joint disease of the shoulder joint complex, having a history of surgical intervention to the shoulder joint complex, having any diagnosed rheumatic, systemic or neurological disease
* Having cardiovascular pathologies that limit rehabilitation

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 20 (Estimated)
Dates: Start 2025-07-28 (Estimated); Primary Completion 2026-09-28 (Estimated); Study Completion 2026-09-28 (Estimated)

PRIMARY OUTCOMES:
Assessment of pain intensity | Change from the initial level after the 6-week treatment program.
  Pain intensity will be assessed with the Visual Analog Scale (VAS). Patients are asked to mark the intensity of pain they feel at rest, during elevation, and at night on the scale. The patient is asked to position the pain intensity between "No Pain at All" and "Very Severe Pain" at one end. The area from the point "0" where there is no pain to the point they mark is measured.
Evaluation of joint range of motion | Change from the initial level after the 6-week treatment program.
  Joint range of motion will be assessed with the smartphone goniometer application. Measurements will be made in the form of painless and painful active joint range of motion and passive joint range of motion assessments of the shoulder in all directions.
Pectoralis minor shortness assessment | Change from the initial level after the 6-week treatment program.
  While standing in a free standing position, the distance between the coracoid process of the scapula and the 4th rib will be measured with a tape measure. The determined length will be divided by the patient's height in cm and multiplied by 100 to obtain the pectoralis minor index (PMI).
Scapular alignment assessment | Change from the initial level after a 6-week treatment program.
  Lateral Scapular Slip Test (LSKT) will be used to assess scapular alignment. It is applied according to the procedure described by Kibler. Accordingly; 3 test positions are used. In the first position; The shoulder glenohumeral joint is in a neutral position, the humerus is in a medial rotation position with 45° abduction in the coronal plane in the second test position, and the shoulder is in a medial rotation position with 90° abduction in the coronal plane in the third test position. In the test where the distance of the scapula from the midline is measured; the horizontal distance from the T4 spinous process to the medial corner of the scapula is measured with a tape measure. A distance difference of 1.5 cm or more between the two sides is defined as positive LSKT by Kibler.
Evaluation of thoracic kyphosis | Change from the baseline after a 6-week treatment program.
  Thoracic kyphosis will be assessed with a smartphone inclinometer application. The short side of the smartphone is placed over the anatomical reference points (T1-T3, T12) marked on the spine. First, the phone is placed on the T1-T3 spinous process and the protractor is set to 0°, then the phone is placed on the T12 spinous process and the angular value displayed on the screen is recorded as the degree of kyphosis.
Evaluation of shoulder-related quality of life | Change from baseline after 6-week treatment program.
  Western Ontario Rotator Cuff Index (WORC): The WORC, whose Turkish adaptation has been shown to be reliable and valid, will be used to determine the effectiveness of rehabilitation on quality of life. It consists of 5 sections including physical symptoms, sports and leisure, work, lifestyle and emotional functions and a total of 21 questions. In the WORC index, evaluation results can be given as raw scores and one hundred points. The best possible score is 0 (% 100) and there is no decrease in the patient's shoulder-related quality of life; the worst possible score is 2100 (% 0) and the patient has a very significant decrease in the shoulder-related quality of life.

CONTACTS AND LOCATIONS:
Overall Officials: Zeynel Abidin Çapa, MSc, Principal Investigator — Hitit University
Locations (1):
- Hitit University, Çorum, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No
Indivudual participant data will be available to the responsible researcher.